CLINICAL TRIAL: NCT07206407
Title: Clinical Trial on Rapid Immune Modulating Effects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 058-010
Record Dates: First submitted 2025-09-10; First posted 2025-10-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Immune Surveillance

STUDY DESIGN:
Intervention Model Description: Double-blinded, placebo-controlled, cross-over study design.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will not be informed on which intervention they consume on a given clinic visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Crossover group 1, randomized (Experimental): Crossover study: Participants consume a test product on each of the two clinic visits, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume the active test product versus placebo over 2 weeks. The order of interventions for this group is A, B.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Nutraceutical blend
- Experimental: Crossover group 2, randomized (Experimental): Crossover study: Participants consume a test product on each of the two clinic visits, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume the active test product versus placebo over 2 weeks. The order of interventions for this group is B, A.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Nutraceutical blend

INTERVENTIONS:
Dietary Supplement: Placebo — Four capsules.
Dietary Supplement: Nutraceutical blend — Four capsules.

SUMMARY:
The goal for this clinical trial is to document rapid effects of a nutritional blend on immune cells. A double-blind, placebo-controlled, cross-over study design will be used.

DETAILED DESCRIPTION:
Clinical trial comparing the acute immune effects of a nutraceutical blend, and a placebo. The nutraceutical blend is based on low molecular weight peptides isolated from cow colostrum ultrafiltrate, mushroom extracts, and vitamin C.

24 subjects will participate in a placebo-controlled, randomized, double-blinded, cross-over study design, wherein they will be consuming placebo or the active nutraceutical blend, separated by a 1-week washout period.

Baseline blood samples are taken 1 hour after participants arrive; the dose is then administered. Additional blood samples are taken 1 hour, 2 hours, and 3 hours following consumption of test product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults;
* Age 18-75 years (inclusive);
* Veins easy to see in one or both arms (to allow for the multiple blood draws);
* Willing to comply with study procedures, including:

  * Maintaining a consistent diet and lifestyle routine throughout the study,
  * Consistent habit of bland breakfasts on days of clinic visits,
  * Abstaining from exercising and nutritional supplements on the morning of a study visit,
  * Abstaining from use of coffee, tea, and soft drinks for at least one hour prior to a clinic visit;
  * Abstaining from music, candy, gum, computer/cell phone use, during clinic visits.

Exclusion Criteria:

* Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery not a problem, including previous removal of appendix and gall bladder);
* Taking anti-inflammatory medications on a daily basis;
* Currently experiencing intense stressful events/ life changes;
* Currently in intensive athletic training (such as marathon runners);
* Currently taking antipsychotic medications such as clozapine, Risperdal, Abilify, Zyprexa or Seroquel;
* An unusual sleep routine (examples: working graveyard shift, irregular routine with frequent late nights, studying, partying);
* Unwilling to maintain a constant intake of supplements over the duration of the study;
* Anxiety about having blood drawn;
* Pregnant, nursing, or trying to become pregnant;
* Known allergies related to ingredients in active test product or placebo.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-28 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Immune cell surveillance | 3 hours after consuming a test product for this study protocol
  Observation of changes in immune cell trafficking, i.e., the changes in immune cell numbers in the peripheral blood following administration. Data is collected as 'cell numbers per uL whole blood' for the following immune cell types:
  * Monocytes
  * NK cells
  * NKT cells
  * T cells
  * non-NK nonT cells

SECONDARY OUTCOMES:
Immune cell activation status | 3 hours after consuming a test product for this study protocol
  Observation of immune cell status of alertness, i.e., the changes in the expression of CD25 and CD69. Data is collected as 'mean fluorescence intensity' for the following immune cell types:
  * Monocytes
  * NK cells
  * NKT cells
  * T cells
  * nonNK nonT cells

CONTACTS AND LOCATIONS:
Overall Officials: Gitte S. Jensen, PhD, Principal Investigator — NIS Labs
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No